CLINICAL TRIAL: NCT00728390
Title: Phase 1 Targeted Combination Trial Of PF-00299804 And CP-751,871 In Patients With Advanced Solid Tumors
Brief Title: A Safety And Efficacy Study Of The Combination Of Oral PF-00299804 And Intravenous CP-751,871 Given Every 3 Weeks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A7471004
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Non-Small Cell; Neoplasm Metastasis
Keywords: advanced cancer refractory advanced non-small cell lung cancer
MeSH Terms: conditions — Carcinoma; Neoplasm Metastasis | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — CP-751,871 at recommended dose on Day 1 and 2 of cycle 1, then on Day 1 every 3 weeks; and PF-00299804 orally at recommended dose once daily.

SUMMARY:
This study will explore the combination of the oral drug PF-00299804 and intravenous CP-751,871 in patients with advanced solid tumor. Each of these drugs have been given separately to patients in prior studies, and this study is to establish the safety and efficacy of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented advanced cancer, Eastern Cooperative Oncology Group (ECOG) 0-1;
* Platelets > 100,000, ANC > 1500;
* Ccr > 60 or serum creat. <1.5
* Non-small cell cancer cohort:
* Eastern Cooperative Oncology Group (ECOG) 0-2, prior platin, < 4 prior chemotherapy regimen
* HgA1C <5.7%

Exclusion Criteria:

* Active Central Nervous System (CNS) metastases;
* prior IGF1-R targeted therapy
* Any history of unstable angina, myocardial infarction or symptomatic congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-12-15 (Actual); Primary Completion 2011-08-09 (Actual); Study Completion 2013-01-29 (Actual)

PRIMARY OUTCOMES:
Overall safety profile characterized by type, frequency, severity (as graded using NCI CTC AE v. 3.0), timing, seriousness and relationship to trial treatment of adverse events and laboratory abnormalities. | 18 months

SECONDARY OUTCOMES:
Plasma Pharmacokinetic Parameters of PF-00299804 and CP-751,871 | 12 months
Progression Free Survival (PFS) | 15 months
Best overall response (OR) defined according to RECIST guidelines. | 12 months
Duration of response (DR) | 15 months
Anti-Drug Antibodies (ADA) response; | 18 months
KRAS mutation and EGFR gene amplification and mutation status in available NSCLC tumor tissue (fresh or archived) (NSCLC MTD Expansion Cohort | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (3):
  - Pfizer Investigational Site, Amherst, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, San Antonio, Texas
- Pfizer Investigational Site, Villejuif, France
- Pfizer Investigational Site, Madrid, Spain

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471004&StudyName=A%20Safety%20And%20Efficacy%20Study%20Of%20The%20Combination%20Of%20Oral%20PF-00299804%20And%20Intravenous%20CP-751%2C871%20Given%20Every%203%20Weeks